CLINICAL TRIAL: NCT05378191
Title: A Phase 2, Comparative, Randomised, Adaptive Trial to Evaluate the Safety and Immunogenicity of One Dose of Comirnaty® in Subjects That Had Received One Dose of Vaxzevria®
Brief Title: Vaccination With COMIRNATY in Subjects With a VAXZEVRIA First Dose
Acronym: CombiVacS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5859; NCT04860739 (obsolete NCT alias)
Record Dates: First submitted 2021-09-21; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Covid19
Keywords: heterologous vaccination
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; CVnCoV COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to immediately receive or not a dose of COMIRNATY in a ratio of 2:1. If primary analysis at 14 days confirms the starting hypothesis, subjects randomized to no vaccination will be considered for administration of one dose of COMINARTY at day 28th according to Public Health Department of the Ministry of Health recommendations on heterologous vaccination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VACCINATION (Active Comparator): One standard dose of COMIRNATY in adult subjects (18 years old) having received prior VAXZEVRIA vaccination.
  Interventions: Drug: COMIRNATY
- NO INTERVENTION (No Intervention): No vaccination in adult subjects (18 years old) having received prior VAXZEVRIA vaccination. If primary analysis at day 14th confirms the starting hypothesis, subjects randomized to this arm will be considered for administration of one dose of COMINARTY at day 28th according to Public Health Department of the Ministry of Health recommendations on heterologous vaccination.

INTERVENTIONS:
Drug: COMIRNATY — One dose of COMIRNATY
  Other Names: COVID-19, mRNA vaccine
  Arms: VACCINATION

SUMMARY:
CombiVacS is a phase 2 randomized, adaptive trial developed to evaluate the immunogenicity of a dose of COMIRNATY after a previous single dose of VAXZEVRIA. A stratification will be made based on the following factors: study site, sex and age. This protocol allows to test the immunogenicity and safety of a heterologous vaccination strategy after a previous single dose of VAXZEVRIA.

DETAILED DESCRIPTION:
This is a randomized, non-blinded, controlled, adaptive, multicenter, Phase II study in subjects aged ≥18 years and in good health or stable clinical situation that have received a previous single dose of VAXZEVRIA. Subjects will be randomized to immediately receive or not a dose of COMIRNATY in a ratio of 2:1. If primary analysis at day 14th confirms the starting hypothesis, subjects randomized to no vaccination will be considered for administration of one dose of COMINARTY at day 28th according to Public Health Department of the Ministry of Health recommendations on heterologous vaccination. In case the primary analysis does not confirm the starting hypothesis, subjects will be followed at the time points defined in the flow-chart without administration of COMIRNATY.

Other heterologous vaccination strategies could be incorporated if deemed necessary for public health reasons. This could include the use of different vaccination strategies including those already marketed vaccines for comparative assessment of their safety and efficacy on SARS-CoV-2 and its variants.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18 years old) having received a prime VAXZEVRIA vaccination between 8 and 12 weeks before the screening visit
* Participants must provide consent indicating that he or she understands the purpose, procedures and potential risks and benefits of the study, and is willing to participate in the study.
* Subjects in good health or stable clinical situation.
* Participant is willing and able to adhere to the procedures specified in this protocol.

Exclusion Criteria:

* Participant has a clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature ≥38.0ºC within 24 hours prior to the planned dose of study vaccine.
* Participant has a known or suspected allergy or history of anaphylaxis or other serious adverse reactions to COMIRNATY excipients.
* Subjects with any contraindication to the administration of COMIRNATY, included pregnancy.
* Subjects with prior documented COVID19 since VAXZEVRIA vaccination.
* Subjects have symptoms or signs compatible with COVID19.
* Subjects participating in a clinical trial in the last three months.
* Any condition or situation precluding or interfering the compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-08-22 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
To assess the humoral immune response against SARS-CoV-2, 14 days after vaccination with COMIRNATY in subjects that received a previous single dose of VAXZEVRIA, as compared with no dosing. | 14 days after randomization
  Antibodies against SARS-CoV-2 spike protein. Measure: BAU/mL

SECONDARY OUTCOMES:
To assess the humoral immune response against SARS-CoV-2, 28 days after vaccination with COMIRNATY in subjects that received a previous single dose of VAXZEVRIA. | 28 days after randomization
  Antibodies against SARS-CoV-2 spike protein. Measure: BAU/mL
To assess the long-term (up to 1 year) humoral immune response against SARS-CoV-2 of a dose of COMIRNATY in subjects that received a previous single dose of VAXZEVRIA. | 3, 6 and 12 months after randomization
  Antibodies against SARS-CoV-2 spike protein (BAU/mL)
To assess the occurrence of symptomatic molecularly confirmed COVID-19 and severity of COVID-19 signs and symptoms after the administration of a dose of COMIRNATY in subjects that received a prior single dose of VAXZEVRIA. | Month 1 - 12
  Number of participants with molecularly confirmed COVID-19 and presence and severity of COVID-19 signs and symptoms as measured by Symptoms of Infection with Coronavirus-19
To evaluate the safety of a dose of COMIRNATY in subjects that received a previous single dose of VAXZEVRIA (solicited adverse events) | Day 1-7
  Number of solicited local and systemic adverse events (AEs) for 7 days after vaccine
To evaluate the safety of a dose of COMIRNATY in subjects that received a previous single dose of VAXZEVRIA (unsolicited adverse events) | Day 1-28
  Number of unsolicited local and systemic adverse events (AEs) for 28 days after vaccine
To evaluate the safety of a dose of COMIRNATY in subjects that received a previous single dose of VAXZEVRIA (serious adverse events) | Month 1-12
  Number of Serious adverse events (SAEs) throughout the study (from randomization until end of the study).
To evaluate the safety of a dose of COMIRNATY in subjects that received a previous single dose of VAXZEVRIA (Medically-attended adverse events) | Month 1-6
  Number of Medically-attended adverse events (MAAEs) from the day of vaccination until 6 months after the last vaccination

OTHER OUTCOMES:
To evaluate the relationship between the immune response measured as NAV (Neutralizing antibodies) and antibodies against SARS-CoV-2 spike protein measured by immunoassay. | Month 1-12
  Neutralizing antibodies (BAU/mL) and antibodies against SARS-CoV-2 spike protein (BAU/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Cristobal Belda Iniesta, MD, PhD, Study Chair — Instituto de Salud Carlos III; Jesús Frías Iniesta, MD, PhD, Principal Investigator — Spanish Clinical Research Network - SCReN; Jose R Arribas, MD, PhD, Study Director — Hospital Universitario La Paz
Locations (5):
- Spain (5):
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Hospital Vall d´Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Will submit data to European Union Drug Regulating Authorities Clinical Trials Database (EudraCT) and share data result.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within one year after study end.
Access Criteria: Published in EudraCT
URL: https://eudract.ema.europa.eu/index.html

REFERENCES:
- [Derived] Garcia-Perez J, Borobia AM, Perez-Olmeda M, Portoles A, Castano L, Campins-Arti M, Bertran MJ, Bermejo M, Arribas JR, Lopez A, Ascaso-Del-Rio A, Arana-Arri E, Fuentes Camps I, Vilella A, Cascajero A, Garcia-Morales MT, Castillo de la Osa M, Perez Ingidua C, Lora D, Jimenez-Santana P, Pino-Rosa S, Gomez de la Camara A, De La Torre-Tarazona E, Calonge E, Cruces R, Belda-Iniesta C, Alcami J, Frias J, Carcas AJ, Diez-Fuertes F; CombiVacS Study Group. Immunogenicity of a third dose with mRNA-vaccines in the ChAdOx1-S/BNT162b2 vaccination regimen against SARS-CoV-2 variants. iScience. 2024 Aug 14;27(9):110728. doi: 10.1016/j.isci.2024.110728. eCollection 2024 Sep 20. PMID 39286494
- [Derived] Garcia-Perez J, Gonzalez-Perez M, Castillo de la Osa M, Borobia AM, Castano L, Bertran MJ, Campins M, Portoles A, Lora D, Bermejo M, Conde P, Hernandez-Gutierrez L, Carcas A, Arana-Arri E, Tortajada M, Fuentes I, Ascaso A, Garcia-Morales MT, Erick de la Torre-Tarazona H, Arribas JR, Imaz-Ayo N, Mellado-Pau E, Agusti A, Perez-Ingidua C, Gomez de la Camara A, Ochando J, Belda-Iniesta C, Frias J, Alcami J, Perez-Olmeda M; CombiVacS study Group. Immunogenic dynamics and SARS-CoV-2 variant neutralisation of the heterologous ChAdOx1-S/BNT162b2 vaccination: Secondary analysis of the randomised CombiVacS study. EClinicalMedicine. 2022 Jul 1;50:101529. doi: 10.1016/j.eclinm.2022.101529. eCollection 2022 Aug. PMID 35795713
- [Derived] Borobia AM, Carcas AJ, Perez-Olmeda M, Castano L, Bertran MJ, Garcia-Perez J, Campins M, Portoles A, Gonzalez-Perez M, Garcia Morales MT, Arana-Arri E, Aldea M, Diez-Fuertes F, Fuentes I, Ascaso A, Lora D, Imaz-Ayo N, Baron-Mira LE, Agusti A, Perez-Ingidua C, Gomez de la Camara A, Arribas JR, Ochando J, Alcami J, Belda-Iniesta C, Frias J; CombiVacS Study Group. Immunogenicity and reactogenicity of BNT162b2 booster in ChAdOx1-S-primed participants (CombiVacS): a multicentre, open-label, randomised, controlled, phase 2 trial. Lancet. 2021 Jul 10;398(10295):121-130. doi: 10.1016/S0140-6736(21)01420-3. Epub 2021 Jun 25. PMID 34181880